CLINICAL TRIAL: NCT01764997
Title: A Randomized, Controlled Study of Sarilumab and Methotrexate (MTX) Versus Etanercept and MTX in Patients With Rheumatoid Arthritis (RA) and an Inadequate Response to 4 Months of Treatment With Adalimumab and MTX
Brief Title: An Evaluation of Sarilumab Plus Methotrexate Compared to Etanercept Plus Methotrexate in RA Patients Not Responding to Adalimumab Plus Methotrexate
Acronym: RA-COMPARE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to small number of participants entering randomization. Not a safety issue.
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC11574; 2012-001984-66; U1111-1131-6653 (Other: UTN)
Record Dates: First submitted 2013-01-08; First posted 2013-01-10 (Estimated); Results first posted 2017-07-27 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — sarilumab; Etanercept; Methotrexate; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Adalimumab Open Label run-in (Experimental): Adalimumab 40 mg every 2 weeks (Q2W) for 16 weeks added to stable dose of MTX.
  Interventions: Drug: Methotrexate; Drug: Adalimumab
- Etanercept + MTX (Randomized) (Active Comparator): Etanercept 50 mg in combination with Placebo for sarilumab Q2W and etanercept 50 mg on alternating weeks for 24 weeks added to stable dose of MTX.
  Interventions: Drug: Etanercept; Drug: Methotrexate; Drug: Placebo (for sarilumab)
- Sarilumab 150 mg + MTX (Randomized) (Experimental): Sarilumab 150 mg in combination with placebo for etanercept Q2W and placebo for etanercept on alternating weeks for 24 weeks added to stable dose of MTX.
  Interventions: Drug: Sarilumab; Drug: Methotrexate; Drug: Placebo (for etanercept)
- Sarilumab 200 mg + MTX (Randomized) (Experimental): Sarilumab 200 mg in combination with placebo for etanercept Q2W and placebo for etanercept on alternating weeks for 24 weeks added to stable dose of MTX.
  Interventions: Drug: Sarilumab; Drug: Methotrexate; Drug: Placebo (for etanercept)
- Sarilumab 150 mg + MTX Open Label Sub-study (Experimental): Sarilumab 150 mg Q2W for 52 weeks added to stable dose of MTX.
  Interventions: Drug: Sarilumab; Drug: Methotrexate

INTERVENTIONS:
Drug: Sarilumab — Pharmaceutical form: Solution for injection in pre-filled syringe; Route of administration: Subcutaneous
  Other Names: SAR153191; REGN88
  Arms: Sarilumab 150 mg + MTX (Randomized); Sarilumab 150 mg + MTX Open Label Sub-study; Sarilumab 200 mg + MTX (Randomized)
Drug: Etanercept — Pharmaceutical form: Solution for injection in pre-filled syringe; Route of administration: Subcutaneous
  Other Names: Enbrel
  Arms: Etanercept + MTX (Randomized)
Drug: Methotrexate — Dispensed according to local practice.
Drug: Placebo (for sarilumab)
  Arms: Etanercept + MTX (Randomized)
Drug: Placebo (for etanercept)
  Arms: Sarilumab 150 mg + MTX (Randomized); Sarilumab 200 mg + MTX (Randomized)
Drug: Adalimumab — Pharmaceutical form: Solution for injection in pre-filled syringe; Route of administration: Subcutaneous
  Arms: Adalimumab Open Label run-in

SUMMARY:
Primary Objective:

To demonstrate the treatment effect of sarilumab and methotrexate (MTX) compared to etanercept and MTX in participants with rheumatoid arthritis (RA) and an inadequate response to adalimumab and MTX by evaluation of the Disease Activity Score for 28 joints (DAS28).

Secondary Objectives:

To assess the signs and symptoms of RA in participants taking sarilumab in combination with MTX.

To assess the quality of life of participants with RA taking sarilumab in combination with MTX.

To assess the safety and tolerability of sarilumab in combination with MTX in participants with RA.

DETAILED DESCRIPTION:
The maximum study duration per participant enrolled in the open label run-in phase and was eligible to enroll in the randomized phase of main study was 54 weeks:

* open label screening period of up to 4 weeks
* open-label treatment period of 16 weeks
* randomized screening period of 2 to 4 weeks
* randomized treatment post-treatment safety follow-up period of 6 weeks.

The maximum study duration per participant enrolled only in the open label run-in phase and was not eligible to enroll in the randomized phase of main study was 26 weeks:

* open label screening period of up to 4 weeks
* open-label treatment period of 16 weeks
* open label treatment post-treatment safety follow-up period of 6 weeks.

The maximum study duration per participant enrolled in the open label run-in phase and was eligible to enroll in the sarilumab sub-study was 82 weeks:

* open label screening period of up to 4 weeks
* open-label treatment period of 16 weeks
* screening period of 2 to 4 weeks
* sarilumab treatment period of 52 weeks
* sub-study post-treatment safety follow-up period of 6 weeks.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of RA >/= 3 months duration.
* Continuous treatment of MTX 10 - 25 mg/week (or per local labeling requirements if the dose range differs) for at least 12 weeks before screening visit and on a stable dose for 8 weeks before screening visit.
* Active disease defined as: at least 6/66 swollen and 8/68 tender joints and high sensitivity C-reactive protein > 10 mg/L.

Exclusion criteria:

* Age < 18 years.
* Use of parenteral corticosteroids or intra-articular corticosteroids within 4 weeks of the screening visit.
* Use of oral corticosteroids in a dose higher than prednisone 10 mg or equivalent per day, or a change in dosage within 4 weeks of the screening visit.
* Prior treatment with a tumor necrosis factor (TNF)-alpha inhibitor, or other biological disease modifying anti-rheumatoid drug (DMARD) or Janus Kinase inhibitor.
* New treatment with or dose-adjustment of on-going nonsteroidal anti-inflammatory drugs (NSAIDs) or cyclo-oxygenase-2 (COX-2) inhibitors within 4 weeks of the screening visit.
* Treatment with traditional oral DMARD /immunosuppressive agents other than MTX within 4 weeks or 12 weeks before the screening visit, depending on DMARD.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 776 (Actual)
Dates: Start 2013-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (257):
- United States (30):
  - Investigational Site Number 840004, Birmingham, Alabama
  - Investigational Site Number 840212, Glendale, California
  - Investigational Site Number 840211, Thousand Oaks, California
  - Investigational Site Number 840049, Upland, California
  - Investigational Site Number 840205, Victorville, California
  - Investigational Site Number 840201, Denver, Colorado
  - Investigational Site Number 840209, Danbury, Connecticut
  - Investigational Site Number 840203, Washington D.C., District of Columbia
  - Investigational Site Number 840210, Clearwater, Florida
  - Investigational Site Number 840128, Ormond Beach, Florida
  - Investigational Site Number 840063, Palm Harbor, Florida
  - Investigational Site Number 840060, Sarasota, Florida
  - Investigational Site Number 840207, Tampa, Florida
  - Investigational Site Number 840018, Idaho Falls, Idaho
  - Investigational Site Number 840213, Indianapolis, Indiana
  - Investigational Site Number 840109, Lake Charles, Louisiana
  - Investigational Site Number 840073, Cumberland, Maryland
  - Investigational Site Number 840202, Hagerstown, Maryland
  - Investigational Site Number 840204, Battle Creek, Michigan
  - Investigational Site Number 840150, Lansing, Michigan
  - Investigational Site Number 840200, Jackson, Mississippi
  - Investigational Site Number 840037, Tupelo, Mississippi
  - Investigational Site Number 840112, Lincoln, Nebraska
  - Investigational Site Number 840056, New York, New York
  - Investigational Site Number 840117, Pittsburgh, Pennsylvania
  - Investigational Site Number 840016, North Charleston, South Carolina
  - Investigational Site Number 840025, Jackson, Tennessee
  - Investigational Site Number 840074, Mesquite, Texas
  - Investigational Site Number 840061, Tacoma, Washington
  - Investigational Site Number 840124, Clarksburg, West Virginia
- Argentina (7):
  - Investigational Site Number 032052, Buenos Aires
  - Investigational Site Number 032050, Buenos Aires
  - Investigational Site Number 032053, La Plata
  - Investigational Site Number 032013, Rosario
  - Investigational Site Number 032005, San Miguel de Tucumán
  - Investigational Site Number 032051, San Miguel de Tucumán
  - Investigational Site Number 032009, Zárate
- Australia (4):
  - Investigational Site Number 036020, Camperdown
  - Investigational Site Number 036004, Heidelberg West
  - Investigational Site Number 036014, Victoria Park
  - Investigational Site Number 036007, Woodville
- Brazil (6):
  - Investigational Site Number 076001, Curitiba
  - Investigational Site Number 076016, Curitiba
  - Investigational Site Number 076006, Goiânia
  - Investigational Site Number 076010, Juiz de Fora
  - Investigational Site Number 076005, Rio de Janeiro
  - Investigational Site Number 076013, Vitória
- Chile (6):
  - Investigational Site Number 152005, Osorno
  - Investigational Site Number 152018, Santiago
  - Investigational Site Number 152001, Santiago
  - Investigational Site Number 152002, Santiago
  - Investigational Site Number 152011, Santiago
  - Investigational Site Number 152015, Temuco
- Colombia (6):
  - Investigational Site Number 170016, Bogotá
  - Investigational Site Number 170040, Bogotá
  - Investigational Site Number 170001, Bogotá
  - Investigational Site Number 170007, Bucaramanga
  - Investigational Site Number 170009, Bucaramanga
  - Investigational Site Number 170041, Medellín
- Czechia (8):
  - Investigational Site Number 203004, Ostrava
  - Investigational Site Number 203032, Prague
  - Investigational Site Number 203001, Prague
  - Investigational Site Number 203031, Prague
  - Investigational Site Number 203033, Prague
  - Investigational Site Number 203030, Prague
  - Investigational Site Number 203002, Uherské Hradiště
  - Investigational Site Number 203006, Zlín
- Ecuador (3):
  - Investigational Site Number 218003, Cuenca
  - Investigational Site Number 218001, Guayaquil
  - Investigational Site Number 218002, Quito
- Finland (5):
  - Investigational Site Number 246001, Helsinki
  - Investigational Site Number 246002, Hyvinkää
  - Investigational Site Number 246030, Oulu
  - Investigational Site Number 246003, Pori
  - Investigational Site Number 246032, Tampere
- France (8):
  - Investigational Site Number 250003, Amiens
  - Investigational Site Number 250007, Bobigny
  - Investigational Site Number 250001, La Roche-sur-Yon
  - Investigational Site Number 250002, Montpellier
  - Investigational Site Number 250005, Paris
  - Investigational Site Number 250004, Paris
  - Investigational Site Number 250006, Strasbourg
  - Investigational Site Number 250008, Toulouse
- Germany (10):
  - Investigational Site Number 276007, Berlin
  - Investigational Site Number 276057, Berlin
  - Investigational Site Number 276058, Cologne
  - Investigational Site Number 276056, Dresden
  - Investigational Site Number 276055, Dresden
  - Investigational Site Number 276051, Erlangen
  - Investigational Site Number 276013, Hamburg
  - Investigational Site Number 276001, Herne
  - Investigational Site Number 276053, Ludwigsfelde
  - Investigational Site Number 276050, Rostock
- Greece (4):
  - Investigational Site Number 300010, Athens
  - Investigational Site Number 300002, Heraklion
  - Investigational Site Number 300014, N. Efkarpia
  - Investigational Site Number 300012, Pátrai
- Hungary (5):
  - Investigational Site Number 348001, Budapest
  - Investigational Site Number 348010, Debrecen
  - Investigational Site Number 348021, Esztergom
  - Investigational Site Number 348013, Gy?r
  - Investigational Site Number 348008, Gyula
- Israel (8):
  - Investigational Site Number 376032, Ashkelon
  - Investigational Site Number 376001, Haifa
  - Investigational Site Number 376010, Haifa
  - Investigational Site Number 376031, Haifa
  - Investigational Site Number 376035, Jerusalem
  - Investigational Site Number 376030, Ramat Gan
  - Investigational Site Number 376011, Tel Aviv
  - Investigational Site Number 376034, Tel Litwinsky
- Italy (5):
  - Investigational Site Number 380002, Florence
  - Investigational Site Number 380004, Genova
  - Investigational Site Number 380005, Genova
  - Investigational Site Number 380041, L’Aquila
  - Investigational Site Number 380042, Valeggio sul Mincio
- Latvia (3):
  - Investigational Site Number 428002, Liepāja
  - Investigational Site Number 428001, Riga
  - Investigational Site Number 428003, Ventspils
- Lithuania (4):
  - Investigational Site Number 440005, Kaunas
  - Investigational Site Number 440006, Klaipėda
  - Investigational Site Number 440010, Panevezys
  - Investigational Site Number 440011, Vilnius
- Malaysia (7):
  - Investigational Site Number 458012, Batu Caves
  - Investigational Site Number 458014, George Town
  - Investigational Site Number 458001, Ipoh
  - Investigational Site Number 458013, Kota Bharu
  - Investigational Site Number 458002, Kuching
  - Investigational Site Number 458010, Malacca
  - Investigational Site Number 458011, Seremban
- Mexico (12):
  - Investigational Site Number 484023, Chihuahua City
  - Investigational Site Number 484027, Ciudad Obregón
  - Investigational Site Number 484029, Deleg. Benito Juárez
  - Investigational Site Number 484013, Guadalajara
  - Investigational Site Number 484018, Guadalajara
  - Investigational Site Number 484010, Mexicali
  - Investigational Site Number 484026, Mexicali
  - Investigational Site Number 484052, Mexico City
  - Investigational Site Number 484004, Mérida
  - Investigational Site Number 484017, México
  - Investigational Site Number 484025, San Luis
  - Investigational Site Number 484051, Tijuana
- New Zealand (4):
  - Investigational Site Number 554007, Auckland
  - Investigational Site Number 554010, Dunedin
  - Investigational Site Number 554005, Hamilton
  - Investigational Site Number 554011, Nelson
- Peru (7):
  - Investigational Site Number 604001, Lima
  - Investigational Site Number 604010, Lima
  - Investigational Site Number 604009, Lima
  - Investigational Site Number 604012, Lima
  - Investigational Site Number 604007, Lima
  - Investigational Site Number 604005, Lima
  - Investigational Site Number 604020, Lima
- Poland (16):
  - Investigational Site Number 616019, Bydgoszcz
  - Investigational Site Number 616054, Bytom
  - Investigational Site Number 616052, Działdowo
  - Investigational Site Number 616015, Elblag
  - Investigational Site Number 616057, Krakow
  - Investigational Site Number 616059, Krakow
  - Investigational Site Number 616061, Krakow
  - Investigational Site Number 616005, Lublin
  - Investigational Site Number 616063, Myślenice
  - Investigational Site Number 616018, Poznan
  - Investigational Site Number 616013, Sosnowiec
  - Investigational Site Number 616056, Starachowice
  - Investigational Site Number 616016, Szczecin
  - Investigational Site Number 616058, Ustroń
  - Investigational Site Number 616051, Warsaw
  - Investigational Site Number 616053, Żyrardów
- Romania (12):
  - Investigational Site Number 642041, Bacau
  - Investigational Site Number 642001, Bucharest
  - Investigational Site Number 642040, Bucharest
  - Investigational Site Number 642002, Bucharest
  - Investigational Site Number 642012, Bucharest
  - Investigational Site Number 642004, Bucharest
  - Investigational Site Number 642023, Bucharest
  - Investigational Site Number 642042, Bucharest
  - Investigational Site Number 642005, Galati
  - Investigational Site Number 642013, Iași
  - Investigational Site Number 642014, Iași
  - Investigational Site Number 642022, Târgovişte
- Russia (16):
  - Investigational Site Number 643006, Kemerovo
  - Investigational Site Number 643056, Krasnoyarsk
  - Investigational Site Number 643052, Moscow
  - Investigational Site Number 643021, Moscow
  - Investigational Site Number 643031, Moscow
  - Investigational Site Number 643030, Moscow
  - Investigational Site Number 643022, Novosibirsk
  - Investigational Site Number 643058, Saint Peterburg
  - Investigational Site Number 643008, Saint Petersburg
  - Investigational Site Number 643010, Samara
  - Investigational Site Number 643011, Saratov
  - Investigational Site Number 643059, Smolensk
  - Investigational Site Number 643013, Ufa
  - Investigational Site Number 643050, Voronezh
  - Investigational Site Number 643057, Yaroslavl
  - Investigational Site Number 643051, Yaroslavl
- South Africa (5):
  - Investigational Site Number 710011, Cape Town
  - Investigational Site Number 710007, Cape Town
  - Investigational Site Number 710008, Pretoria
  - Investigational Site Number 710006, Pretoria
  - Investigational Site Number 710010, Stellenbsoch
- South Korea (11):
  - Investigational Site Number 410020, Busan
  - Investigational Site Number 410006, Busan
  - Investigational Site Number 410013, Daegu
  - Investigational Site Number 410005, Daejeon
  - Investigational Site Number 410011, Jeonju
  - Investigational Site Number 410016, Seoul
  - Investigational Site Number 410015, Seoul
  - Investigational Site Number 410022, Seoul
  - Investigational Site Number 410023, Seoul
  - Investigational Site Number 410021, Seoul
  - Investigational Site Number 410008, Suwon
- Spain (8):
  - Investigational Site Number 724009, A Coruña
  - Investigational Site Number 724043, Córdoba
  - Investigational Site Number 724042, Madrid
  - Investigational Site Number 724041, Madrid
  - Investigational Site Number 724040, Madrid
  - Investigational Site Number 724001, Málaga
  - Investigational Site Number 724011, Sabadell
  - Investigational Site Number 724012, Santiago de Compostela
- Taiwan (5):
  - Investigational Site Number 158010, Changhua
  - Investigational Site Number 158004, Chiayi City
  - Investigational Site Number 158012, Kaohsiung City
  - Investigational Site Number 158011, Kaohsiung City
  - Investigational Site Number 158006, Taipei
- Thailand (4):
  - Investigational Site Number 764002, Bangkok
  - Investigational Site Number 764010, Bangkok
  - Investigational Site Number 764003, Bangkok Noi
  - Investigational Site Number 764011, Khon Kaen
- Ukraine (21):
  - Investigational Site Number 804003, Dnipropetrovsk
  - Investigational Site Number 804002, Donetsk
  - Investigational Site Number 804024, Donetsk
  - Investigational Site Number 804029, Ivano-Frankivsk
  - Investigational Site Number 804010, Kharkiv
  - Investigational Site Number 804001, Kharkiv
  - Investigational Site Number 804025, Kiev
  - Investigational Site Number 804023, Kyiv
  - Investigational Site Number 804014, Kyiv
  - Investigational Site Number 804027, Kyiv
  - Investigational Site Number 804011, Kyiv
  - Investigational Site Number 804030, Lutsk
  - Investigational Site Number 804005, Lviv
  - Investigational Site Number 804033, Lviv
  - Investigational Site Number 804020, Lviv
  - Investigational Site Number 804032, Odesa
  - Investigational Site Number 804022, Odesa
  - Investigational Site Number 804012, Odesa
  - Investigational Site Number 804021, Simferopol
  - Investigational Site Number 804028, Zaporizhzhya
  - Investigational Site Number 804031, Zhytomyr
- United Kingdom (7):
  - Investigational Site Number 826023, Barnsley
  - Investigational Site Number 826022, Birmingham
  - Investigational Site Number 826021, Dudley
  - Investigational Site Number 826026, Durham
  - Investigational Site Number 826027, Durham
  - Investigational Site Number 826020, Harlow
  - Investigational Site Number 826025, Wigan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 228 sites in 31 countries. A total of 1949 participants were screened between 09 May 2013 and 07 Aug 2014 of which 1173 participants were screen failures and a total of 776 participants entered in the adalimumab run-in phase of the study.
Pre-assignment Details: Of 776 participants, 365 completed adalimumab run-in phase, of whom 43 non-responders randomized (1:1:1) in double-blind fashion to receive sarilumab 150 mg, sarilumab 200 mg or etanercept 50 mg; 322 responders entered in open label sub-study. 373 participants did not proceed into randomized phase or sub-study and 38 discontinued from run-in phase.
Groups:
- Adalimumab Open Label run-in: Adalimumab 40 mg subcutaneous (SC) injection every 2 weeks (Q2W) for 16 weeks added to stable dose of methotrexate (MTX).
- Etanercept + MTX (Randomized): Etanercept 50 mg SC injection in combination with Placebo for sarilumab Q2W and etanercept 50 mg SC injection on alternating weeks for 24 weeks added to stable dose of MTX.
- Sarilumab 150 mg + MTX (Randomized): Sarilumab 150 mg SC injection in combination with placebo for etanercept Q2W and placebo for etanercept on alternating weeks for 24 weeks added to stable dose of MTX.
- Sarilumab 200 mg + MTX (Randomized): Sarilumab 200 mg SC injection in combination with placebo for etanercept Q2W and placebo for etanercept on alternating weeks for 24 weeks added to stable dose of MTX.
- Sarilumab 150 mg + MTX Open Label Sub-study: Sarilumab 150 mg SC injection Q2W for 52 weeks added to stable dose of MTX.
Period: Run-in Period
Arm/Group | Adalimumab Open Label run-in | Etanercept + MTX (Randomized) | Sarilumab 150 mg + MTX (Randomized) | Sarilumab 200 mg + MTX (Randomized) | Sarilumab 150 mg + MTX Open Label Sub-study
Started | 776 | 0 | 0 | 0 | 0
Completed | 738 (43 participants proceeded to randomized treatment and 322 proceeded to open-label sub-study.) | 0 | 0 | 0 | 0
Not Completed | 38 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 15 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 5 | 0 | 0 | 0 | 0
Not completed — Poor compliance to protocol | 1 | 0 | 0 | 0 | 0
Not completed — Other than specified above | 17 | 0 | 0 | 0 | 0
Period: Study Drug Treatment Period
Arm/Group | Adalimumab Open Label run-in | Etanercept + MTX (Randomized) | Sarilumab 150 mg + MTX (Randomized) | Sarilumab 200 mg + MTX (Randomized) | Sarilumab 150 mg + MTX Open Label Sub-study
Started | 0 | 17 | 13 | 13 | 322
Completed | 0 | 16 | 13 | 13 | 286
Not Completed | 0 | 1 | 0 | 0 | 36
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 24
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 2
Not completed — Other than specified above | 0 | 0 | 0 | 0 | 10

BASELINE CHARACTERISTICS:
Population: All participants who included in open label run-in period, randomized treatment and sub-study.
Groups:
- Adalimumab Open Label run-in Treatment Only: Adalimumab 40 mg SC injection Q2W for 16 weeks added to stable dose of MTX during run-in period. Participants who were not randomized in the main study or did not enter the sub-study were included in this arm for safety assessment.
- Total: Total of all reporting groups
Arm/Group | Adalimumab Open Label run-in Treatment Only | Etanercept + MTX (Randomized) | Sarilumab 150 mg + MTX (Randomized) | Sarilumab 200 mg + MTX (Randomized) | Sarilumab 150 mg + MTX Open Label Sub-study | Total
Number analyzed (Participants) | 411 | 17 | 13 | 13 | 322 | 776
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 360 | 14 | 10 | 10 | 274 | 668
  >=65 years | 51 | 3 | 3 | 3 | 48 | 108
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 342 | 15 | 10 | 9 | 261 | 637
  Male | 69 | 2 | 3 | 4 | 61 | 139

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Disease Activity Score for 28 Joints - C-Reactive Protein (DAS28-CRP) Score at Week 24
Time Frame: Baseline, Week 24
Population: As the number of participants randomized fell well below target (43 vs. 699), the efficacy data were not systematically collected or cleaned and no datasets have been created to report.
Arm/Group | Etanercept + MTX (Randomized) | Sarilumab 150 mg + MTX (Randomized) | Sarilumab 200 mg + MTX (Randomized)
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With at Least 20% Improvement in American College of Rheumatology (ACR20), at Least 50% Improvement in ACR (ACR50) and at Least 70% Improvement in ACR (ACR70) Efficacy Response Rates at Week 12 and Week 24
Time Frame: Week 12 and Week 24
Population: as for outcome 1
Arm/Group | Etanercept + MTX (Randomized) | Sarilumab 150 mg + MTX (Randomized) | Sarilumab 200 mg + MTX (Randomized)
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Percentage of Participants Achieving Clinical Remission Score (DAS28-CRP) <2.6 at Week 12 and Week 24
Time Frame: Week 12 and Week 24
Population: as for outcome 1
Arm/Group | Etanercept + MTX (Randomized) | Sarilumab 150 mg + MTX (Randomized) | Sarilumab 200 mg + MTX (Randomized)
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Change From Baseline in DAS28-CRP Score at Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 1
Arm/Group | Etanercept + MTX (Randomized) | Sarilumab 150 mg + MTX (Randomized) | Sarilumab 200 mg + MTX (Randomized)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to the final visit (Week 16 for run-in period and Week 58 for treatment period) regardless of seriousness or relationship to investigational product
Description: Reported AEs are treatment-emergent AEs that is AEs that developed/worsened during the 'on-treatment period' (the time from the first dose of adalimumab to the end of follow-up period). All participants who entered open-label run-in period were included for safety assessment.
Groups:
- Adalimumab Open Label run-in: Adalimumab 40 mg SC injection Q2W for 16 weeks added to stable dose of MTX. AEs in this group were those collected from signature of the informed consent form up to the end of Adalimumab treatment (Week 16).
- Etanercept + MTX (Randomized): Etanercept 50 mg SC injection in combination with Placebo for sarilumab Q2W and etanercept 50 mg SC injection on alternating weeks for 24 weeks added to stable dose of MTX. AEs in this group were those collected post randomization up to the final visit (Week 30).
- Sarilumab 150 mg + MTX (Randomized): Sarilumab 150 mg SC injection in combination with placebo for etanercept Q2W and placebo for etanercept on alternating weeks for 24 weeks added to stable dose of MTX. AEs in this group were those collected post randomization up to the final visit (Week 30).
- Sarilumab 200 mg + MTX (Randomized): Sarilumab 200 mg SC injection in combination with placebo for etanercept Q2W and placebo for etanercept on alternating weeks for 24 weeks added to stable dose of MTX. AEs in this group were those collected post randomization up to the final visit (Week 30).
- Sarilumab 150 mg + MTX Open Label Sub-study: Sarilumab 150 mg SC injection Q2W for 52 weeks added to stable dose of MTX. AEs in this group were those collected from enrollment in the sub-study up to the final visit (Week 58).
Arm/Group | Adalimumab Open Label run-in | Etanercept + MTX (Randomized) | Sarilumab 150 mg + MTX (Randomized) | Sarilumab 200 mg + MTX (Randomized) | Sarilumab 150 mg + MTX Open Label Sub-study
Serious Adverse Events (participants affected / at risk) | 25/776 | 2/17 | 0/13 | 0/13 | 11/322
Other Adverse Events (participants affected / at risk) | 132/776 | 7/17 | 7/13 | 8/13 | 104/322
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab Open Label run-in (N=776) | Etanercept + MTX (Randomized) (N=17) | Sarilumab 150 mg + MTX (Randomized) (N=13) | Sarilumab 200 mg + MTX (Randomized) (N=13) | Sarilumab 150 mg + MTX Open Label Sub-study (N=322)
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Cholecystitis infective (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Colonic abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Escherichia pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Histoplasmosis disseminated (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Tuberculous pleurisy (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Viral parotitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Blindness (Eye disorders) | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Ischaemia (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Gastroduodenitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Influenza B virus test positive (Investigations) | 1 | 0 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0 | 0 | 0
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab Open Label run-in (N=776) | Etanercept + MTX (Randomized) (N=17) | Sarilumab 150 mg + MTX (Randomized) (N=13) | Sarilumab 200 mg + MTX (Randomized) (N=13) | Sarilumab 150 mg + MTX Open Label Sub-study (N=322)
Body tinea (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Hordeolum (Infections and infestations) | 2 | 0 | 1 | 0 | 0
Onychomycosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 7 | 0 | 0 | 1 | 3
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Rash pustular (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 7 | 0 | 0 | 1 | 5
Tinea versicolour (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 27 | 1 | 1 | 1 | 16
Urinary tract infection (Infections and infestations) | 16 | 1 | 0 | 0 | 4
Viral pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 1 | 2 | 33
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 10 | 0 | 0 | 1 | 5
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 8 | 1 | 0 | 1 | 3
Tooth disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 4 | 1 | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 1 | 0 | 0 | 4
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 2
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 2
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 0 | 0 | 1 | 2
Injection site erythema (General disorders) | 9 | 0 | 0 | 1 | 15
Injection site pain (General disorders) | 9 | 0 | 0 | 1 | 3
Injection site pruritus (General disorders) | 5 | 1 | 0 | 0 | 9
Injection site rash (General disorders) | 6 | 0 | 1 | 1 | 7
Injection site swelling (General disorders) | 0 | 0 | 0 | 1 | 2
Peripheral swelling (General disorders) | 1 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 7 | 0 | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 5 | 0 | 0 | 2 | 11
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 1 | 3
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 4
Accidental overdose (Injury, poisoning and procedural complications) | 24 | 0 | 3 | 0 | 14
Chillblains (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was prematurely terminated due to small number of participants entering randomization.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.